CLINICAL TRIAL: NCT02851160
Title: Perceptions and Representations of Cancer Chemotherapy
Acronym: chemotherapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL16_0208
Record Dates: First submitted 2016-06-30; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2015-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Psycho-Oncology

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients requiring lung cancer chemotherapy: 30 major Patients with lung cancer requiring chemotherapy either as palliative or adjuvant as surgical treatment having a semi-structured interview conducted by a clinical psychologist
  Interventions: Other: semi-structured interview conducted by a clinical psychologist
- Family of lung cancer patients receiving chemotherapy: 30 Family of lung cancer patients receiving chemotherapy having a semi-structured interview conducted by a clinical psychologist
  Interventions: Other: semi-structured interview conducted by a clinical psychologist
- doctors caring for lung cancer patients receiving chemotherapy: 15 doctors caring for lung cancer patients receiving chemotherapy 15 have a semi-structured interview conducted by a psychiatrist specialized in psycho-oncology
  Interventions: Other: semi-structured interview conducted by a psychiatrist specialized in psycho-oncology

INTERVENTIONS:
Other: semi-structured interview conducted by a clinical psychologist — semi-structured interview conducted by a clinical psychologist
  Groups: Family of lung cancer patients receiving chemotherapy; Patients requiring lung cancer chemotherapy
Other: semi-structured interview conducted by a psychiatrist specialized in psycho-oncology — semi-structured interview conducted by a psychiatrist specialized in psycho-oncology
  Groups: doctors caring for lung cancer patients receiving chemotherapy

SUMMARY:
Qualitative study on data from interviews such patients, relatives and doctors involved in the implementation of cancer care. Framework type of method using grounded theory

DETAILED DESCRIPTION:
The word chemotherapy itself, because it belongs to the secular knowledge and therefore Doxa is a hard word, which stores what it is stable, common and therefore impersonal. It has the properties of a symbol, that is to say that joint several meanings, some of which are contradictory.

The objective of the research:

To determine the perceptions and representations of chemotherapy, its physical impacts, psychological and relational.

To qualitatively compare the performances of chemotherapy as it has an end as scheduled for adjuvant chemotherapy, or endless precise as in the palliative chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* 30 major Patients with lung cancer requiring chemotherapy either as palliative or adjuvant as surgical treatment
* 30 significant others (relatives) major applicant lung cancer patients chemotherapy either palliation or as adjuvant to surgery
* 15 Doctors oncologists performing either chemotherapy as palliative or adjuvant as surgical treatment

Exclusion Criteria:

* NA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 30 major Patients with lung cancer requiring chemotherapy either as palliative or adjuvant as surgical treatment
  * 30 significant others (relatives) major applicant lung cancer patients chemotherapy either palliation or as adjuvant to surgery
  * 15 Doctors oncologists performing either chemotherapy as palliative or adjuvant as surgical treatment
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The semi-structured interview | 1 day (day of inclusion)
  The interview will be analyzed in a framework type of method (grounded theory) in accordance with the guidelines coreq.

IPD SHARING:
Plan to Share IPD: Undecided